CLINICAL TRIAL: NCT02941003
Title: Establishment and Evaluation for Pathological Diagnostic Criteria of Intraoperative Frozen Section of Early Stage Lung Cancer
Brief Title: Precision Diagnosis for Intraoperative Frozen Section of Early Stage Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jie Zhang, Chief Physician, Shanghai Chest Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: Chest005
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Lung Cancer
Keywords: Early stage lung adenocarcinoma; Intraoperative frozen section; Diagnostic criteria
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OCT treatment (Experimental): Randomly assigned patients whose small pulmonary nodules are inflated with the diluted OCT medium (2:3) used for frozen section, and then detected under microscope for their histopathological characteristics, by immunostaining for specific protein expression, by NGS (next-generation sequencing) for driver mutations.
  Interventions: Device: microscope; Other: immunostaining; Device: NGS
- OCT free (Experimental): Randomly assigned patients whose small pulmonary nodules are uninflated with OCT used for frozen section, and then detected under microscope for their histopathological characteristics, by immunostaining for specific protein expression, by NGS for driver mutations.
  Interventions: Device: microscope; Other: immunostaining; Device: NGS

INTERVENTIONS:
Device: microscope — Detection of of histopathological characteristics of OCT treatment or OCT free samples from patients .
Other: immunostaining — Detection of CD31/CD34, D2-40, Ki67 and p53 immunostaining of OCT treatment or OCT free samples from patients .
Device: NGS — The investigators used the device to detect the gene mutations of OCT treatment or OCT free samples obtained from part of the patients.
  Other Names: Illumina Nexseq500

SUMMARY:
The purpose of this study is:

1. To establish a set of diagnostic criteria of intraoperative frozen section of early stage lung adenocarcinoma, including clinicopathologic and molecular characteristics.
2. To assess its clinical usefulness in guiding surgical procedure for early stage lung adenocarcinoma.

DETAILED DESCRIPTION:
The detection rate of small pulmonary nodules is increasing due to the widespread use of high-resolution computed tomography (CT) screening in clinical practice. These minute pulmonary nodules are suggestive of atypical adenomatous hyperplasia (AHH), adenocarcinoma in situ (AIS), minimally invasive adenocarcinoma (MIA), and invasive adenocarcinoma. Hence, the precision diagnosis of intraoperative frozen section is particularly imperative for its fundamental role in assess indeterminate lung lesions and guide the extent of subsequent surgical procedure.

However, it is still difficult for the surgical pathologist to apply the various features according to the newly revised WHO classification of lung adenocarcinoma (2015) to guide surgical management due to their unascertained accuracy or heterogeneity of lung cancer or technique problem. Therefore, the establishment and assessment for a set of diagnostic criteria of intraoperative frozen section of early stage lung adenocarcinoma are our primary aim in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with suspected pulmonary nodules (5~20 mm) by chest CT scan;
2. Patients received surgical operation.

Exclusion Criteria:

1. Patients compliance is poor and cannot accept follow-up;
2. Patients nursing or pregnant;
3. Patients with a history of any cancer;
4. Patients with confirmed pathological diagnosis or received radiotherapy or chemotherapy or target therapy preoperatively.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-12 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of histopathological characteristics between intraoperative frozen section and paraffin section for patients with early stage lung adenocarcinoma | 6 months

SECONDARY OUTCOMES:
Detection of CD31/CD34, D2-40, Ki67 and p53 among different subtypes of early stage lung adenocarcinoma by immunohistochemical (IHC) analysis | 6 months
Comparison of mutation profiles among different subtypes of early stage lung adenocarcinoma by tissue microdissection and subsequent next generation sequencing (NGS) | 6 months
Verification of the driver mutations from NGS results using droplet digital PCR (ddPCR) in early stage lung adenocarcinoma. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jie Zhang, MD, MS., Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided